CLINICAL TRIAL: NCT01210898
Title: A Phase IIIB, Observer-Blind, Randomized, Parallel Groups, Extension Study to Evaluate the Immunogenicity and Safety Following a Single Intramuscular Dose of a Sub-unit Adjuvanted or a Non-adjuvanted Influenza Vaccines in Healthy Children Previously Vaccinated in the V70P5 Study
Brief Title: Immunogenicity and Safety of V70P5 Revaccination Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V70P5E1; 2010-021644-18 (EudraCT Number)
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2012-01

CONDITIONS: Influenza
Keywords: Influenza; Trivalent; Adjuvanted; Vaccine; Children
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (13):
- Group 1 (Experimental)
  Interventions: Biological: Adjuvanted seasonal influenza vaccine
- Group 2 (Experimental)
  Interventions: Biological: Adjuvanted seasonal influenza vaccine
- Group 3 (Experimental)
  Interventions: Biological: Adjuvanted seasonal influenza vaccine
- Group 4 (Experimental)
  Interventions: Biological: Adjuvanted seasonal influenza vaccine
- Group 5 (Experimental)
  Interventions: Biological: Adjuvanted seasonal influenza vaccine
- Group 6 (Experimental)
  Interventions: Biological: Adjuvanted seasonal influenza vaccine
- Group 7 (Experimental)
  Interventions: Biological: Adjuvanted seasonal influenza vaccine
- Group 8 (Experimental)
  Interventions: Biological: Adjuvanted seasonal influenza vaccine
- Group 9 (Experimental)
  Interventions: Biological: Adjuvanted seasonal influenza vaccine
- Group 10 (Experimental)
  Interventions: Biological: Adjuvanted seasonal influenza vaccine
- Group 11 (Experimental)
  Interventions: Biological: Adjuvanted seasonal influenza vaccine
- Group 12 (Experimental)
  Interventions: Biological: Adjuvanted seasonal influenza vaccine
- Group 13 (Experimental)
  Interventions: Biological: Adjuvanted seasonal influenza vaccine

INTERVENTIONS:
Biological: Adjuvanted seasonal influenza vaccine — Full or half dose of adjuvanted seasonal influenza vaccine; Full or half dose of unadjuvanted seasonal influenza vaccine

SUMMARY:
This study will evaluate the safety and immunogenicity of children previously primed in the V70P5 study when revaccinated with adjuvanted or unadjuvanted seasonal influenza vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female children that have previously participated in the V70P5 study in Finland.

Exclusion Criteria:

* Any condition which in the opinion of the investigator may interfere with the evaluation of the study objectives.

Ages: 18 Months to 96 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 197 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Evaluate immunogenicity of children primed and revaccinated with adjuvanted influenza vaccine by GMR, seroprotection | 22 days post vaccination
Evaluate immunogenicity of children primed and revaccinated with a half dose of adjuvanted influenza vaccine by GMR, Seroprotection and seroconversion | 22 days post vaccination
Evaluate immunogenicity of children primed with adjuvanted influenza vaccine and revaccinated with unadjuvanted influenza vaccine by GMR, Seroprotection and seroconversion | 22 days post vaccination
Safety and tolerability of a single dose of adjuvanted or unadjuvanted influenza vaccine stratified according to previous influenza vaccine received | 22 days post vaccination

SECONDARY OUTCOMES:
Primary immunogenicity outcomes as per CBER criteria | Day 22
Compare Immunogenicity of each randomization arm by GMT, GMR, seroconversion and seroprotection by Homologous and Heterologous strains | Day 22

CONTACTS AND LOCATIONS:
Locations (16):
- Finland (16):
  - University of Tampere Medical School, Vaccine Research Center / Tampere yliopisto rokotetutkimuskeskus, Biokatu 10, Tampere
  - Helsinki South, Vaccine Research Clinic, Vuorikatu 18, 3 floor, Helsinki
  - Helsinki East, Vaccine Research Clinic, Itäkeskuksen kauppakeskus/Agenttitalo, Turunlinnantie 8, 4.floor, Helsinki
  - Järvenpää, Vaccine Research Clinic, Yhteiskouluntie 17, Jarvenpaa
  - Kokkola Vaccine Research Clinic, Rantakatu 7, Kokkola
  - Kotka Vaccine Research Clinic, Karjalantie 10-12, Kotka
  - Kuopio Vaccine Research Clinic, Microkatu 1, N-building, 2nd floor, PL 1188, Kuopio
  - Lahti Vaccine Research Clinic, Vesijärvenkatu 74, Lahti
  - Oulu Vaccine Research Clinic, Kiviharjunlenkki 6, Oulu
  - Pori Vaccine Research Clinic, Yrjönkatu 23 (4th floor), Pori
  - Seinäjoki Vaccine Research Clinic, Keskuskatu 6, Seinäjoki
  - Tampere Vaccine Research Clinic, Pinninkatu 47 (1. floor), Tampere
  - Espoo Vaccine Research Clinic, Länsituulentie 10, 4th floor, Tapiontori 1, Espoo
  - Turku Vaccine Research Clinic, Lemminkäisenkatu 14-18 B (4th floor), Turku
  - Vantaa East, Vaccine Research Clinic, Asematie 11 a 16, Vantaa
  - Vantaa West, Vaccine Research Clinic, Jönsaksentie 6 B, 3rd floor, Vantaa

REFERENCES:
- [Result] Vesikari T, Forsten A, Arora A, Tsai T, Clemens R. Influenza vaccination in children primed with MF59-adjuvanted or non-adjuvanted seasonal influenza vaccine. Hum Vaccin Immunother. 2015;11(8):2102-12. doi: 10.1080/21645515.2015.1044167. PMID 26091244